CLINICAL TRIAL: NCT06614062
Title: Clinical Study of 18F Labeled Probe Targeting Fibroblast Activation Protein Inhibitor and Integrin Avβ3 (FAPI-RGD) in Ovarian Cancer,comparison with 18F-FDG
Brief Title: Clinical Study of 18F-FAPI-RGD in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH-Ovarian cancer
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Observational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the value of 18F-FAPI-RGD PET/CT imaging in ovarian cancer. Participants will undergo clinical evaluation and 18F-FAPI-RGD PET/CT examination and compare it with 18F-FDG PET/CT imaging.

DETAILED DESCRIPTION:
Ovarian cancer is the malignant tumor with the highest mortality rate among women, and also the most intractable gynecological malignant tumor in clinical treatment. Its incidence rate and mortality are increasing year by year. China's incidence rate of ovarian cancer ranks first in the world.Due to the lack of typical clinical symptoms and effective screening tools in the early stage, more than 70% of patients were in advanced cancer when diagnosed,that is, there was peritoneal and/or distant metastasis. The mortality rate was high (mortality/incidence rate ratio was 60%) , the radical cure rate was low, and the 5-year overall survival rate was only 30% . The survival rate of ovarian cancer is closely related to staging (stage I 5-year survival rate is 92%, stage IV is 5%) . Therefore, early and accurate detection and staging are of great significance for the selection of treatment methods and the improvement of patient survival rate.Positron emission tomography (PET) is a non-invasive molecular imaging technique. Currently, 18F-FDG PET/CT has been included as a routine examination in the postoperative evaluation of the NCCN ovarian cancer diagnosis and treatment guidelines as a supplementary examination method for preoperative evaluation. Therefore, 18F-FDG PET/CT is recommended by NCCN as an imaging biomarker for ovarian cancer, and performs well in early diagnosis, treatment planning, and postoperative evaluation. However, FDG PET/CT also has some limitations, such as its sensitivity being influenced by different histological subtypes (such as ovarian mucinous carcinoma, clear cell carcinoma, or low-grade serous carcinoma). In addition, false negatives caused by physiological high uptake in the intestine and false positives caused by ovarian physiological uptake and some benign lesions (such as cystadenoma, endometrioma, and acute inflammatory processes) still exist. Therefore, a more effective imaging technique is needed to improve the detection and staging of ovarian tumors.

α V β 3-Integrins play a crucial role in promoting and maintaining angiogenesis, and have been identified as biomarkers of angiogenesis. Research has found that integrins α V β 3 is highly expressed in neovascular endothelial cells and tumor cells, including ovarian cancer, and plays an important role in regulating tumor growth, angiogenesis, local invasion, and metastasis potential.Research has shown that 68 Ga-FAPI-04 is a novel radioligand targeting fibroblast activating protein (FAP), which has recently been used for tumor microenvironment imaging, especially cancer associated fibroblasts (CAFs), with promising imaging results . Research has shown that compared to 18F-FDG, 68Ga-FAPI PET/CT has higher sensitivity in detecting and diagnosing lymph node and peritoneal metastases in ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:• Age 18 and above• Patients who have been diagnosed with, or are clinically highly suspected of, Ovarian cancer and have had no other treatment within 3 months -

Exclusion Criteria:• Patients with a second primary tumor• Pregnant or breastfeeding• Severe liver or kidney disease•Claustrophobia or other PET/CT scan contraindications

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed or highly suspected Ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Correlation between clincal indicater and PET/CT results | 2 months
  Correlation of ultrasound, CT, tumor markers and 18F-FAPI-RGD PET/CT results。

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Nuclear Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No